CLINICAL TRIAL: NCT06741553
Title: A Study That Uses an Organized System to Prospectively Collect Uniform Data From a Defined Population
Brief Title: Prospective Cohort Study of Patients With Early Alzheimer's Disease Treated With Lecanemab
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1113; 82371190 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-11-29; First posted 2024-12-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment (MCI)
Keywords: Alzheimer Disease; Lecanemab; Cognition; Amyloid-related imaging abnormalities
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — lecanemab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — All study subjects underwent blood collection before the 1st dose (V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39) for routine blood tests, liver and kidney function, plasma biomarkers, and other indicators. Among them, the APOE genotype of subjects will be tested before the 1st dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Treated Group: This is an observational study. The investigators included early AD patients treated with Lecanemab, and evaluated them by plasma, magnetic resonance imaging (MRI) examination and clinical scale. The investigators observed the changes in MRI characteristics and clinical symptoms of patients after Lecanemab administration, evaluated the improvement effect of Lecanemab on cognitive function, and monitored the risk factors of adverse reactions.
  Interventions: Drug: Lecanemab 10 mg/kg

INTERVENTIONS:
Drug: Lecanemab 10 mg/kg — Lecanemab was administered 10mg/kg every two weeks.

SUMMARY:
As the population increases and aging intensifies, cognitive disorders represented by Alzheimer's disease (AD) not only pose a severe threat to public health but also bring significant social and economic burdens. Previously, treatment options for Alzheimer's disease were very limited, mainly providing symptomatic relief with few available medications. Lecanemab, an FDA-approved clinical treatment drug in 2023, targets the core pathology of AD-abnormal amyloid-beta (Aβ) aggregation in the brain-and has been validated through both biomarker and clinical scale assessments. The optimal dosage and safety-efficacy profile of lecanemab for treating early AD have been observed in phase 2 and phase 3 clinical trials. However, the use of lecanemab may lead to certain adverse effects, including infusion-related reactions, amyloid-related imaging abnormalities (ARIA), such as microhemorrhages or hemosiderin deposits (ARIA-H), and ARIA-E. This study aims to establish a prospective follow-up cohort of patients treated with lecanemab to observe changes in cranial imaging characteristics and clinical symptoms, assess the cognitive improvement effects of lecanemab in early AD patients (stages 3-4), and monitor the risk factors for adverse event occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination (MMSE) score between 22 and 30, Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) score between 0.5 and 1;
* Confirmation of positive amyloid pathology by Amyloid-PET or cerebrospinal fluid Aβ testing;
* Completion of APOE gene testing.
* Willingness to use Lecanemab.

Exclusion Criteria:

* Unable to tolerate MRI scans;
* MRI showing hemorrhagic manifestations, including >4 microbleeds, surface iron deposition in any region, previous major hemorrhage, or potential brain lesions or vascular malformations;
* Use of anticoagulants or antiplatelet drugs, presence of hemorrhagic diseases, or any other conditions that increase the risk of central nervous system bleeding;
* With unstable physical conditions, unstable mental disorders, or those who are pregnant or breastfeeding.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included early AD patients treated with Lecanemab at the Second Affiliated Hospital of Zhejiang University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
CDR-SB Score | CDR-SB scales by baseline before the 1st dose(V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39)
  All study subjects underwent Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) assessment by a specialist before the 1st dose (V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39). CDR-SB, with total scores ranging from 0 to 18, can be used to measure cognitive changes in the early stages of Alzheimer's disease, with higher scores indicating more severe symptoms.
MMSE | MMSE scales by baseline before the 1st dose(V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39)
  All study subjects underwent Mini Mental State Examination (MMSE) assessment by a specialist before the 1st dose (V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39). MMSE, with total scores ranging from 0 to 30, can be used to measure cognitive changes in the early stages of Alzheimer's disease, with lower scores indicating more severe symptoms.
ADCs-ADL | ADCs-ADL scales by baseline before the 1st dose(V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39)
  All study subjects underwent Alzheimer's Disease Cooperative Study-Activity of Daily Life (ADCs-ADL) assessment by a specialist before the 1st dose (V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39). CDR-SB, with total scores ranging from 0 to 78, can be used to measure activity of daily life changes in the early stages of Alzheimer's disease, with lower scores indicating more severe symptoms.
NPI | NPI scales by baseline before the 1st dose(V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39)
  All study subjects underwent Neuropsychiatric Inventory (NPI) assessment by a specialist before the 1st dose (V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39). CDR-SB, with total scores ranging from 0 to 18, can be used to measure cognitive changes in the early stages of Alzheimer's disease, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Aβ-PET Burden | Aβ-PET tested by baseline before the 1st dose(V1) , at 12 and 18 months after treatment (V25,V39)
  All study subjects underwent Aβ positron emission tomography (PET) before the 1st dose (V1) ,at 12 and 18 months after treatment (V26,V39). The investigators quantified participants' Aβ burden using the average cortical standard uptake value ratio (SUVR), that is, tracer uptake in medial orbital frontal, lateral temporal, parietal, anterior cingulate, posterior cingulate, and precuneus regions divided by uptake in the cerebellar reference region.
MRI | Time Frame: MRI tested by baseline before the 1st dose(V1) , at 2, 3, 6, 12 and 18 months after treatment (V5, V7, V14, V25, V39)
  All study subjects underwent magnetic resonance imaging (MRI) before the 1st dose (V1) ,at 2, 3, 6,12 and 18 months after treatment. The scan includes T1, T2 fluid attenuated inversion recovery (FLAIR, 5 mm slice thickness), susceptibility weighted imaging (SWI, 1 mm slice thickness) and diffusion weighted imaging (DWI). The MRI scan can be used to meature the study subjects' hippocampus atrophy and white matter hyperintensities and to detect whether adverse events such as amyloid-related imaging abnormalities happen.
Biospecimen | Blood tested by baseline before the 1st dose(V1) , at 3, 6,12 and 18 months after treatment(V7, V14, V25, V39)
  All study subjects underwent blood collection before the 1st dose (V1) and at 3, 6, 12, and 18 months after treatment (V7, V14, V25, V39) for routine blood tests, liver and kidney function, plasma biomarkers, and other indicators. Among them, the APOE genotype of subjects will be tested before the 1st dose.

CONTACTS AND LOCATIONS:
Overall Officials: Baorong Zhang, M.D., Study Director — Zhejiang University School of Medicine Second Affiliated Hospital
Locations (1):
- Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No